CLINICAL TRIAL: NCT03607734
Title: Penicillin Allergy De-Labelling in Elective Surgical Patients - A Study to Determine the Safety, Efficacy and Feasibility of Abbreviated Allergy Testing
Brief Title: Penicillin Allergy De-Labelling in Elective Surgical Patients (PADLES)
Acronym: PADLES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AN17/92982
Record Dates: First submitted 2018-06-27; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Amoxicillin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 - Interventional Treatment (Other): A graded oral challenge test, using amoxicillin in syrup form, will be administered as follows:
  * 50mg amoxicillin (10% total dose)
  * 250mg amoxicillin (50% total dose)
  * 200mg amoxicillin (remainder needed to complete a 500mg full dose) A 20 minute interval will separate each dose given, and participants will be observed throughout the test. They will be required to stay for one hour after the final dose has been administered. Fully trained staff and all equipment for emergency resuscitation will be immediately available.
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — A graded oral challenge test, using amoxicillin in syrup form, will be administered as follows:
  * 50mg amoxicillin (10% total dose)
  * 250mg amoxicillin (50% total dose)
  * 200mg amoxicillin (remainder needed to complete a 500mg full dose) A 20 minute interval will separate each dose given, and participants will be observed throughout the test. They will be required to stay for one hour after the final dose has been administered. Fully trained staff and all equipment for emergency resuscitation will be immediately available.

SUMMARY:
Penicillin antibiotics are safe and inexpensive, and target selected bacteria rather than killing a broad range. Unfortunately, around 10% of the population are labelled as 'penicillin allergic'. This is often based on side effects such as rash and diarrhoea, and 90-95% of people with the label are not actually allergic to the drug.

The label leads to the use of alternative antibiotics, which tend to more toxic, and less specific about which bacteria they kill; this increases the risk of infections with so-called 'super-bugs', compared to patients without the label. People with the label also have an increased length of hospital stay and rates of readmission. These are significant problems for individuals, as well as wider society. Where the diagnosis is in doubt, the gold standard test for allergy is an oral challenge. Patients undergo skin +/- blood tests prior to a challenge, as these can help make the diagnosis. This combined pathway is expensive and time consuming, so testing cannot be offered routinely to all patients. However in patients with 'historic' reactions (many years previously), skin and blood tests become much less useful; in one study, 100% of patients who skin tested positive for amoxycillin allergy, tested negative 5 years later. Patients with historic reactions can therefore proceed directly to an oral challenge without prior skin or blood testing, since these offer little help in making the diagnosis. This streamlines the pathway, making it quick, non-invasive and cheap. Already established practice in several centres in Europe and beyond, this abbreviated pathway is offered on an ad-hoc basis in some centres in the UK.

The aim is to demonstrate that this pathway offers a safe and effective way to perform large-scale delabelling of elective surgical patients, who might not otherwise meet NICE criteria for testing.

ELIGIBILITY:
Inclusion Criteria:

* Allergic history is historic (more than 10 years ago) and suggestive of a non-immediate reaction or side effect
* Requires penicillin as first-line treatment for their planned surgery
* >18 years
* Willing and able to give consent

Exclusion Criteria:

* Not willing to participate
* History suggestive of immediate type reaction (anaphylaxis)
* History of toxic epidermal necrolysis or Stevens Johnson syndrome
* Pregnant, planning to become pregnant during study, or breastfeeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Completion of the study questionnaire by participants | 1 day
  Online questionnaire about previously diagnosed allergies to be completed by study participants

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No